CLINICAL TRIAL: NCT03894189
Title: The Effect of Doxapram Versus Theophylline on Diaphragmatic Function and Weaning From Mechanical Ventilation After Open Heart Surgery
Brief Title: The Effect of Doxapram Versus Theophylline on Diaphragmatic Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Samaa Abou Alkassem Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Faculty Of Medicine,Beni -Suef
Record Dates: First submitted 2019-03-23; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Weaning Failure
MeSH Terms: interventions — Doxapram; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- doxapram group (GROUP D) (Active Comparator): The patients in this group will receive loading dose of (1 mg/kg) followed by an infusion of (1mg/kg/h)
  Interventions: Drug: Doxapram Hydrochloride; Drug: Theophylline
- theophylline group (GROUP T) (Active Comparator): the therapeutic loading dose (5mg/kg) followed by an infusion of (0.5 mg/kg/h)
  Interventions: Drug: Doxapram Hydrochloride; Drug: Theophylline

INTERVENTIONS:
Drug: Doxapram Hydrochloride — the diaphragmatic function will be assessed measuring right and left diaphragmatic thickening fraction in the two groups to be compared as a primary outcome using ultrasound. following the administration of the selected drug
  Other Names: Doxapram
Drug: Theophylline — the diaphragmatic function will be assessed measuring right and left diaphragmatic thickening fraction in the two groups to be compared as a primary outcome using ultrasound. following the administration of the selected drug

SUMMARY:
Doxapram is licensed for drug-induced post-anesthesia respiratory depression , arousal effect and return airway protective reflexes caused by barbiturates, volatile anesthetics, nitrous oxide or benzodiazepines over dosage.

Value of theophylline to stimulate the respiratory neuronal network has been examined by previous studies and increases the activity of respiratory muscles, including the intercostal , transversus abdominis muscles and the diaphragm, it also has bronchodilator and anti-inflammatory effects.

DETAILED DESCRIPTION:
This randomized comparative study will be conducted in the post-surgical cardio-thoracic intensive care unit in Beni -Suef University Hospital after approval of the department of anesthesiology, surgical ICU and pain management , and cardio thoracic department and the local ethics and research committee, and obtaining written informed consents from the patients to compare the effect of doxapram versus theophylline on diaphragmatic function using ultrasonography parameter: thickening fraction of the diaphragmatic muscle during respiration which defined as [(thickness at end-inspiration - thickness at end-expiration)/thickness at end-expiration] during spontaneous breathing trial as a primary outcome and its effect on weaning time and weaning success rate as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria: Patients (males and females) in the age group 20 -60 scheduled for elective open heart surgery ( e.g. coronary artery bypass grafting, valve replacement ) under cardiopulmonary bypass .

-

Exclusion Criteria:The preoperative exclusion criteria:

1. Age older than 60 years
2. Preoperative left ventricular ejection fraction less than 30%
3. Chronic obstructive pulmonary disease
4. Significant hepatic disease (alanine aminotransferase or aspartate aminotransferase >150 U/l).
5. Renal failure (creatinine >200 μm).
6. History of seizure, or stroke.
7. History of diaphragmatic palsy, cervical spine injury, or neuromuscular disease (eg, myasthenia gravis, Guillain-Barré syndrome).
8. Lesion adjacent to the diaphragm
9. Intra-abdominal hypertension (intra-abdominal pressure ≥12 mm Hg )
10. Known allergy to the study drugs.

The Post enrollment exclusion criteria:

1. Postoperative hemorrhage (chest tube drainage ≥ 200 ml/h).
2. Surgical complications necessitating reoperation.
3. Postoperative cardiac failure necessitating high-dose inotropes or intra -aortic balloon pump.
4. Refractory hypoxemia (ratio of arterial oxygen tension [PaO2] to fraction of inspired oxygen [FIO2] <150 mmHg).
5. Occurrence of neurologic deficit.
6. -Myocardial ischemia (ST-segment depression) lasting more than 30 min
7. Failure of spontaneous breathing trial.

   -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the effect of doxapram versus theophylline on diaphragmatic function | the study drugs will be infused for 1 hour,At the end of 60 min of SBT, the diaphragmatic function will be assessed measuring right and left diaphragmatic thickening fraction in the two groups to be compared as a primary outcome using ultrasound.
  : thickening fraction of the diaphragmatic muscle during respiration which defined as [(thickness at end-inspiration - thickness at end-expiration)/thickness at end-expiration](18) (19) during spontaneous breathing trial as a primary outcome and its effect on weaning time and weaning success rate as secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Samaa ak Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt